CLINICAL TRIAL: NCT01340157
Title: Randomized, Open Study to Assess the Impact of Two Different Types of Food on the Relative Bioavailability of Fexinidazole Tablets After Single Oral Dose in Healthy Male Volunteers
Brief Title: Fexinidazole (1200mg) Bioavailability Under Different Food Intake Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Antoine Tarral, MD, Drugs for Neglected Diseases Initiative
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DNDiFEX002
Record Dates: First submitted 2011-04-14; First posted 2011-04-22 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2011-04

CONDITIONS: PK in Healthy Volunteers
Keywords: Fexinidazole; Phase I; Bioavailability study; Food effect; Human African Trypanosomiasis
MeSH Terms: interventions — fexinidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fasting (Experimental): Treatment A: 1200mg fexinidazole administered in fasting conditions by oral route
  Interventions: Drug: Fexinidazole
- Meal 1: Plumpy Nuts (Experimental): Treatment B: 1200mg fexinidazole administered in fed conditions (meal 1) by oral route
  Interventions: Drug: Fexinidazole
- Meal 2: Rice + beans (Experimental): Treatment B: 1200mg fexinidazole administered in fed conditions (meal 2) by oral route
  Interventions: Drug: Fexinidazole

INTERVENTIONS:
Drug: Fexinidazole — Single oral dose of 1200mg fexinidazole consisting of 2 tablets dosed at 600mg per tablet.

SUMMARY:
The present study is designed to assess the impact of concomitant food intake on the relative bioavailability of a single oral fexinidazole tablet administration.

ELIGIBILITY:
Inclusion Criteria:

* Male healthy volunteers 18 to 45 years of age,
* All subjects to be of sub-Saharan African origins with both parents of sub- Saharan African origins too,
* Male subjects with a body mass index (BMI) calculated as weight in kg/(height in m2) from 18 to 28 kg/m2 at screening,
* Able to communicate well with the Investigator and research staff and to comply with the requirements of the entire study,
* Provision of written informed consent to participate as shown by a signature on the volunteer consent form,
* Light smokers (less than 10 cigarettes per day) or subjects who are non-smokers. No smoking (or use of smoking substitute e.g. nicotine patch) is permitted from screening throughout the study,
* Normal arterial blood pressure (BP) and pulse rate or, if abnormal, considered not clinically significant by the principal Investigator. These will be measured after resting for 5 min,
* Registered with the French Social Security in agreement with the French law on biomedical experimentation.

Exclusion Criteria:

* Who on direct questioning and physical examination have evidence of any clinically significant acute or chronic disease, including known or suspected Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection,
* With any clinically significant abnormality following review of pre-study laboratory tests (aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT) and alkaline phosphatase (ALP) must be within normal ranges), vital signs, full physical examination and Electrocardiogram (ECG),
* Who are within the exclusion period defined in the National Register for Healthy Volunteers of the French Ministry of Health,
* Who forfeit their freedom by administrative or legal award or who were under guardianship,
* Unwilling to give their informed consent,
* Who have a positive laboratory test for Hepatitis B surface antigen (HbsAg), or anti-HIV 1/2 or anti- HCV antibodies
* Who have a history of allergy, intolerance or photosensitivity to any drug,
* Who have a history of serious allergy, asthma, allergic skin rash or sensitivity to any drug,
* Who are known or suspected alcohol or drug abusers (more than 14 units of alcohol per week, one unit = 8 g or about 10 mL of pure alcohol),
* Who drink more than 8 cups daily of beverage containing caffeine,
* Who have a positive laboratory test for urine drug screening (opiates, cocaine, amphetamine, cannabis, benzodiazepines),
* Who have undergone surgery or have donated blood within 12 weeks prior to the start of the study,
* Who have taken any prescribed or over the counter drug (including antacid drug), with the exception of paracetamol (up to 3 g per day) within 2 weeks prior to the first dose administration,
* Who have any clinical condition or prior therapy which, in the opinion of the Investigator, made the subject unsuitable for the study,
* Who participated to any clinical trial with an investigational drug in the past 3 months preceding study entry.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Plasma concentration measurement of fexinidazole, fexinidazole sulfoxide and sulfone metabolites after a single oral dose of fexinidazole (1200mg) administration and under different food intake conditions

SECONDARY OUTCOMES:
Occurence of AEs
  To assess safety and tolerability of fexinidazole tablets administered as single oral dose under fasting conditions and after two different meals in healthy male volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Hovsepian, MD, Principal Investigator — SGS Aster; Antoine Tarral, MD, Study Director — Drugs for Neglected Diseases initiative
Locations (1):
- SGS Aster s.a.s., Paris, France

REFERENCES:
- See also: Sponsor website — http://www.dndi.org
- See also: Publication combining results of NCT00982904 & NCT01483170 — http://www.dndi.org/wp-content/uploads/2009/06/ClinicalPK_Tarral_FexinidazoleHAT_2014.pdf